CLINICAL TRIAL: NCT01542372
Title: Two Stepped Care Models for PTSD Among Cambodian Refugees With PTSD
Brief Title: Two Stepped Care Models for Posttraumatic Stress Disorder (PTSD) Among Cambodian Refugees With PTSD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inadequate flow of patients
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Devon E. Hinton, Associate Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH094312
Record Dates: First submitted 2012-02-21; First posted 2012-03-02 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: PTSD; Cognitive behavioral therapy (CBT); Medication augmentation; Treatment-resistant PTSD; Cambodian refugees; Culturally sensitive treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Medication augmentation (Active Comparator): In one arm, the patients will be given a medication augmentation for SSRI/SSRN-resistant PTSD
  Interventions: Drug: Medication augmentation
- CBT augmentation (Active Comparator): In this arm, patients will receive CBT to treat SSRI/SSRN-resistant PTSD.
  Interventions: Behavioral: CBT

INTERVENTIONS:
Drug: Medication augmentation
  Other Names: Prazosin is the first choice agent in this Arm
  Arms: Medication augmentation
Behavioral: CBT
  Other Names: Cognitive-Behavioral Therapy
  Arms: CBT augmentation

SUMMARY:
This project aims to investigate the efficacy of two models to treat Posttraumatic Stress Disorder (PTSD) for Cambodian refugees in primary care. The first step in both models is giving a medication, which is a serotonin reuptake inhibitor/serotonin-norepinephrine reuptake inhibitor (SSRI/SSRN), with paroxetine being the first-line agent. For those patients who still have PTSD, the second step is either another medication or a culturally sensitive cognitive behavioral therapy (CBT). The investigators hypothesize that patients will improve in both models, but more so in the the CBT model.

DETAILED DESCRIPTION:
This project aims to investigate the efficacy of two models to treat PTSD for Cambodian refugees in primary care. The first step in both models is giving a medication (an SSRI/SSRN, e.g., paroxetine). For those who still have PTSD, the second step is either adding another medication (e.g., prazosin) or providing culturally sensitive cognitive behavioral therapy (CBT). We hypothesize that patients will improve in both models, but more so in the the CBT model. The primary outcome measure is PTSD severity as assessed by the PTSD Checklist (PCL). Eligibility requirements include having PTSD and having been old enough to remember the Khmer Rouge period.

ELIGIBILITY:
Inclusion Criteria:

* PTSD;
* PCL great or equal to 44;
* Survivor of the Cambodian genocide;
* At least 7 years old at the time of the Cambodian genocide

Exclusion Criteria:

* Pregnant;
* Active suicidality;
* Mental retardation;
* Organic mental disorder;
* Bipolar disorder;
* Alcohol dependence;
* Marijuana dependence;
* Unable to give conformed consent

Min Age: 43 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Devon E. Hinton, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in primary care clinics
Pre-assignment Details: In Step 1 of the protocol, patients were given an SSRI/SSRN to determine eligibility for Step 2. If a patient still had PTSD (PCL > 30) after Step I, the patient was assigned to an arm of Step 2, which was Medication or CBT augmentation. Of 114 patients started in Step I, 22 met criteria for entry to Step 2, the study proper, addressing study aims.
Groups:
- Medication Augmentation (Prazosin): In this arm, the patients were given a medication augmentation for SSRI/SSRN-resistant PTSD, with the preferred first-line agent being prazosin.
  Prazosin as first-line agent: Prazosin .5 to 2 mg
- CBT Augmentation: In this arm, patients were given CBT to treat SSRI/SSRN-resistant PTSD.
  Cognitive Behavioral Therapy for PTSD: This is a culturally sensitive CBT for the treatment of PTSD
Period: Overall Study
Arm/Group | Medication Augmentation (Prazosin) | CBT Augmentation
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients who meet inclusion criteria for Step 1 such as PTSD and impairment.
Groups:
- Step I: SSRI/SSRN Treatment of PTSD: At Step I, patients receive an SSRI or SSRN to treat PTSD. If a treatment course of SSRI/SSRN does not reduce PTSD to indicated levels, then the patient enters Step 2, which has two arms: Medication or CBT augmentation
Arm/Group | Step I: SSRI/SSRN Treatment of PTSD
Number analyzed (Participants) | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 114
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 44
Region of Enrollment [Number; unit: participants]
  United States | 114

OUTCOME MEASURES:

1. Primary Outcome: Change in the PTSD Checklist (PCL) at 12 Weeks in Step II
Description: A measure of PTSD severity, which is the PTSD Checklist. Total score range is 17 to 85, with a higher score indicating greater psychopathology. Change scores were calculated.
Time Frame: Baseline and 12 weeks
Population: Patients with PTSD checklist scores of 30 or above were eligible for Step II, which was medication augmentation or CBT augmentation.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Medication Augmentation (Prazosin); CBT Augmentation: At Step I, patients receive an SSRI or SSRN to treat PTSD. If a treatment course of SSRI/SSRN does not reduce PTSD to indicated levels, then the patient enters Step 2, which has two arms: Medication or CBT augmentation
Arm/Group | Medication Augmentation (Prazosin) | CBT Augmentation
Number analyzed (Participants) | 11 | 11
units on a scale | -5.0 (9.6) | -11.4 (7.5)

2. Secondary Outcome: Change in the HSCL Anxiety Scale at 12 Weeks in Step II
Description: A measure of anxiety severity, which is the HSCL Anxiety Scale. Each item is rated on a 1-4 Likert-type scale, with a higher score indicating worse psychopathology. Mean scale scores were used, giving a minimum of 1 and a maximum of 4. Change scores were calculated.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medication Augmentation (Prazosin) | CBT Augmentation
Number analyzed (Participants) | 11 | 11
units on a scale | -0.4 (0.6) | -0.6 (0.9)

3. Secondary Outcome: Change in the HSCL Depression Scale at 12 Weeks in Step II
Description: A measure of depression severity, which is the HSCL Depression Scale. Each item is rated on a 1-4 Likert-type scale, with a higher score indicating worse psychopathology. Mean scale scores were used, giving a minimum of 1 and a maximum of 4. Change scores were calculated.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medication Augmentation (Prazosin) | CBT Augmentation
Number analyzed (Participants) | 11 | 11
units on a scale | -0.3 (0.7) | -0.5 (0.7)

4. Secondary Outcome: Change in the SCL Anger Severity at 12 Weeks in Step II
Description: A measure of anger severity, which is the SCL Anger Scale. Each item is rated on a 0-4 Likert-type scale, with a higher score indicating worse psychopathology. Mean scale scores were used, giving a minimum of 0 and a maximum of 4. Change scores were calculated.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medication Augmentation (Prazosin) | CBT Augmentation
Number analyzed (Participants) | 11 | 11
units on a scale | -0.3 (0.8) | -0.9 (0.7)

5. Secondary Outcome: Change in the Cambodian Culturally Sensitive Complaint Profile at 12 Weeks in Step II
Description: A measure of somatic symptoms and cultural syndromes commonly found among distressed Cambodian refugees. Each item is rated on a 0-4 Likert-type scale, with a higher score indicating worse psychopathology. Mean scale scores were used, giving a minimum of 0 and a maximum of 4. Change scores were calculated.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medication Augmentation (Prazosin) | CBT Augmentation
Number analyzed (Participants) | 11 | 11
units on a scale | -0.5 (0.6) | -0.9 (0.5)

6. Secondary Outcome: Change in the SF-12 at 12 Weeks in Step II
Description: A measure of severity of self-perceived functioning. Total score ranges from 0 to 100, with a higher score indicating better self-perceived functioning. Change scores were calculated.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medication Augmentation (Prazosin) | CBT Augmentation
Number analyzed (Participants) | 11 | 11
units on a scale | 6.8 (9.3) | 10.2 (9.0)

ADVERSE EVENTS:
Time Frame: 1 year 7 months
Description: We followed the clinical trials definitions.
Groups:
- Step I and Step 2: Step 1 is treatment with SSRI or SSRN. Step 2 is Medication or CBT augmentation.
Arm/Group | Step I and Step 2
All-Cause Mortality (participants affected / at risk) | 0/114
Serious Adverse Events (participants affected / at risk) | 0/114
Other Adverse Events (participants affected / at risk) | 0/114

LIMITATIONS AND CAVEATS:
Owing to lack of recruitment sites the study was ended early. In addition, many more patients than anticipated had no PTSD after Step I and hence could not be randomized to participate in Step II. This greatly impacted on flow.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No